CLINICAL TRIAL: NCT02727868
Title: Assessment of the Mutation of Pig-A Gene as Biomarker of Genotoxic Exposure in Humans
Acronym: PIG-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-42; 2015-A01753-46 (Registry Identifier: ID RCB)
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Patient With Breast Cancer
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exclusive breast irradiation group (Other): to assess the impact of irradiation areas
  Interventions: Genetic: blood samples
- breast and sternal irradiation group (Other): to assess the impact of irradiation areas
  Interventions: Genetic: blood samples

INTERVENTIONS:
Genetic: blood samples

SUMMARY:
The evaluation of the impact of environment on the incidence of cancer is a major public health issue. Increased knowledge in this area is necessary for the implementation of primary prevention means with appropriate preventive measures but also to the implementation of secondary prevention measures with targeted screening actions.

Among the environmental exposures that may lead to cancer, mutagenic environments are of major importance, and the causal link between environmental genotoxicity and cancer has been established for a long time. It is also well established that susceptibility to mutation is highly variable among individuals. This is explained by genetic polymorphisms of genes involved in metabolism and in genome stability.

The identification of biomarkers of exposure to mutagenic environments is necessary for assessing the impact of an environment in humans. Some studies in animals have shown that the PIG-A gene may be a biomarker of exposure to a mutagenic environment. In particular, a significant increase in erythrocyte PIG-A mutants has been demonstrated in rats after a genotoxic exposure to cisplatin, but it has so far not been evaluated in humans. One study of healthy volunteers shows that the frequency of PIG-A mutated cells in humans can be estimated efficiently and reliably.

The PIG-A gene meets all the necessary criteria for a sentinel gene for tracking of spontaneous somatic mutation frequency or induced a mutagenic environment: ubiquitous expression, phenotypic change linked to a mono-allelic mutation viability of mutated cells , spectrum off inactivating mutations (deletions, substitutions, chromosomal rearrangements). Finally, the detection of the disappearance of glycosylphosphatidylinositol on the plasma membrane is easily achievable by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Major patients,
* The patients achieving a breast cancer
* Patients who have benefited from a breast surgery
* Patients to have an external adjuvant radiotherapy.
* Patients being able to read and understand French.
* Patients beneficiaries of a social security scheme.
* Pregnant women can not participate in this study. A pregnancy test should only be prescribed when clinically indicated, regardless of the course of the study.
* Patients who received information and signed informed consent

Exclusion Criteria:

Patients who received chemotherapy before radiation therapy.

* Minor patients
* Patients who do not speak French and / or unable to read and understand French.
* Patients who have had radiotherapy history
* Patients who have had a history of chemotherapy
* Patients who have not received the information and had not signed informed consent for participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
analysis of the frequency of granulocytes PIG-A mutated | 24 months
  The analyzes will be applied at T0 to determine the intra-assay reproducibility. The frequency distributions of mutated cells will be compared:
  * Between the two groups of patients at T0 then,
  * Within each group between T0 (before exposure), T1 (in process), T2 (end of treatment) and T3 (in therapeutic monitoring post) using non-parametric tests on paired and unpaired.
analysis of the binucleated cell micronuclei frequency in culture | 24 months
  Determining the frequency of micronucleated binucleate cells in culture will be performed on the samples at T0 and T3 each patient of both groups. The frequency distribution of micronucleated cells will be compared within each group between T0 and T3 using non-parametric tests on paired series.
  A difference shall be considered significant if p <0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided